CLINICAL TRIAL: NCT05756933
Title: Noninvasive and Continuous Arterial Waveform Analysis for Predicting Post-induction Hypotension of Endoscopic Surgery Patients.
Brief Title: Arterial Waveform Analysis for Predicting Post-induction Hypotension
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: MOST 111-2221-E-038-019
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-02

CONDITIONS: Hypotension on Induction
Keywords: Anesthesia induction; hypotension; pressure waveform; machine learning
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to develop a computation model for accurately predicting post-induction hypotension in patients receiving laparoscopic surgery under general anesthesia. The main question[s] it aims to answer are:

• whether the corresponding characteristics on pressure wave forms could be use to predict post-induction hypotension.

Participants will be observed before and after induction of general anesthesia for non-invasive arterial pressure wave forms and blood pressure changes.

DETAILED DESCRIPTION:
In this project, an equivalent circuit model will firstly be established to simulate patient's hemodynamics. This model will be applied into analyzing blood pressure wave forms in the MIMIC II database. It will facilitate deep understanding of the effects of induction drugs on pressure waveforms. As a result, the corresponding characteristics on pressure wave forms will be identified. The extracted characteristics from the MIMIC II database will then be applied for developing a computation model via machining learning approaches. The developed model will be validated with another available dataset of 100 patients. This project will then conduct a non-invasive and observational clinical study of 50 patients to prove the clinical value of this project. In this trial, a novel pressure sensor will be employed on patient's fingertip to continuously collect pressure waveform before and after anesthesia induction. Medical records and vital signs will also be collected for exploring the potential of the developed model for predicting other events. Endoscopic surgery patients will be recruited in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 20 years
* Ease of access to the hand used for the ArteVu device during the one-hour it is being used during the operation.
* Able to provide written informed consent for participation in the study.

Exclusion Criteria:

* Pregnant patients.
* Medical or surgical condition that prevents the ability to apply the ArteVu device on an upper extremity finger for a period of one-hour during anesthesia and operation.
* Impaired skin integrity of the fingers (e.g. injuries to the finger, burn injuries, or skin graft surgery on the finger).
* Operations involving the upper extremities or the blood vessels of the upper extremities.
* Arthritis or severe deformities of the hand and fingers
* Prosthetic devices or jewelry (such as a wedding band) that cannot be removed from the finger to be used for the ArteVu device.
* History of malignant hyperthermia
* Raynaud's disease affecting the fingers or hands.
* Topical allergy to ABS or silicone
* Swelling, edema or lymphedema of the upper extremity
* Participants with upper extremity occlusive peripheral vascular diseases
* Inability of the patient to provide written informed consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving laparoscopic surgeries under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
waveform characteristics predicting post-induction hypotension | Evaluated during the induction period of general anesthesia.
  An equivalent circuit model will firstly be established to simulate patient's hemodynamics. This model will be applied into analyzing blood pressure waveforms in the MIMIC II database.

SECONDARY OUTCOMES:
effects of induction effects of induction drugs on vessels | off-line analysis
  Evaluate the specific effects of anesthetics on characteristics of pressure waveform.

CONTACTS AND LOCATIONS:
Overall Officials: Chuen-Chau Chang, MD, PhD, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Department of Anesthesia, Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No